CLINICAL TRIAL: NCT03265509
Title: Assessment of the Effect of Glutamine Supplementation in Addition to Exercise on Pelvic Floor Muscle Strength and Clinical Parameters in Women With Urinary Incontinence or Pelvic Organ Prolapse
Brief Title: Effect of Glutamine on Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Gulistan Bahat-Ozturk, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/1203
Record Dates: First submitted 2017-08-26; First posted 2017-08-29 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutamine (Active Comparator): 30 g/day Glutamine supplementation for three months
  Interventions: Dietary Supplement: glutamine supplementation
- Fantomalt (Placebo Comparator): 30 g/day Fantomalt supplementation for three months
  Interventions: Dietary Supplement: fantomalt supplementation

INTERVENTIONS:
Dietary Supplement: glutamine supplementation — 30 g/day glutamine supplementation for three months
  Arms: Glutamine
Dietary Supplement: fantomalt supplementation — 30 g/day fantomalt supplementation for three months
  Arms: Fantomalt

SUMMARY:
The objective of this study is to determine to effect of additional oral glutamine to Kegel exercises on pelvic floor strength and clinical parameters of urinary incontinence in females with either urinary incontinence (stress and/or urgency) and pelvic prolapse.

DETAILED DESCRIPTION:
Urinary incontinence is a prevalent and costly condition that affects approximately 38% of older community-dwelling women (age>60 years). Incontinence predisposes patients to other health problems, contributes to depression and social isolation, is a significant source of dependency among the elderly, and is widely cited as a factor in nursing home admissions. Sarcopenia is age-related and is characterized by loss of muscle mass, strength and endurance. There is not only a decrease in the number of muscle fibers, but also atrophy in the remaining ones. Several studies indicate glutamine supplementations lead to better muscle performance by stimulate muscle producing in extremities. Similarly, we assume glutamine supplementation could increase pelvic muscle mass and improve the pelvic floor strength. From this point, using glutamine supplementation may effect positively on stress, urge or mixed incontinence, and pelvic prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Presence of urinary incontinence and/or pelvic prolapse and/or decreased vaginal muscle strength in gynaecological examination

Exclusion Criteria:

* Uncontrolled diabetes
* Cognitive dysfunction hampering participation in exercise or assessment

Ages: 45 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle strength with dynamometer | 3 months
  vaginal dynamometer
Pelvic floor muscle strength with digital palpation | 3 months
  digital vaginal palpation method

SECONDARY OUTCOMES:
body composition | 3 months
  muscle mass assessed by bioimpedance analysis
quality of life related prolapse | 3 months
  Prolapse quality of life (PQOL) questionnaire
general quality of life | 3 months
  King's Health Questionnaire (KHQ)
24 hour pad test | 3 months
  assessment of the severity of urinary incontinence as determined by the 24-hour pad weight
hand grip strength | 3 months
  Jamar hand dynamometer
urinary incontinence dairy | 3 months
  urinary incontinence dairy
degree of prolapse | 3 months
  systematic pelvic examination

CONTACTS AND LOCATIONS:
Overall Officials: Gulistan Bahat Ozturk, Ass. Prof., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No